CLINICAL TRIAL: NCT05397600
Title: Efficacy and Safety Assessment of T4032 (Unpreserved Bimatoprost 0.01%) Versus Lumigan® 0.01% in Ocular Hypertensive or Glaucomatous Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT4032-302
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2023-11

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- T4032 (Experimental)
  Interventions: Drug: Bimatoprost Ophthalmic
- Lumigan (Active Comparator)
  Interventions: Drug: Bimatoprost Ophthalmic

INTERVENTIONS:
Drug: Bimatoprost Ophthalmic — Eyedrops

SUMMARY:
The main study purpose is to demonstrate the non-inferiority of T4032 compared to Lumigan® 0.01% in terms of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent dated and signed.
* Both eyes diagnosed open-angle glaucoma or ocular hypertension

Exclusion Criteria:

* History of trauma, infection, clinically significant inflammation within the previous 3 months
* Known or suspected hypersensitivity to one of the components of the Investigational Medicinal Product(s)
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Day 1) to Week 2, Week 6, and Week 12 in IOP. | up to Week12
  Change from baseline (Day 1) to Week 2, Week 6, and Week 12 in IOP at three time points (8:00 a.m.; 10:00 a.m.; 4:00 p.m.) in the study eye.

CONTACTS AND LOCATIONS:
Locations (63):
- United States (55):
  - Arizona Eye Center - Chandler, Chandler, Arizona
  - Eye Physicians & Surgeons of Arizona - Glendale Office, Glendale, Arizona
  - Arizona Glaucoma Specialists - Phoenix, Phoenix, Arizona
  - Walman Eye Center - Sun City, Sun City, Arizona
  - Velvet Clinical Research, Burbank, California
  - Specialty Eye Care Medical Center - Glendale, Glendale, California
  - Global Research Management, Inc., Glendale, California
  - Inland Eye Specialists - Hemet, Hemet, California
  - Diabetic Eye Medical Clinic - Inglewood, Inglewood, California
  - Lakeside Vision Center - Irvine, Irvine, California
  - Sage Eyecare, Los Angeles, California
  - Global Vision Eye Care - Los Angeles- Rock Central, Los Angeles, California
  - North Valley Eye Medical Group, Inc., Mission Hills, California
  - California Eye Specialists Medical Group Inc. - Monrovia, Monrovia, California
  - Aesthetic Eye Care Institute - Eye Research Foundation, Newport Beach, California
  - Foothill Eye Institute - Pasadena, Pasadena, California
  - North Bay Eye Associates - Petaluma - 104 Lynch Creek Way, Petaluma, California
  - California Eye Specialists Medical Group Inc. - Redlands, Redlands, California
  - OC Surgical Eye Institute, Santa Ana, California
  - Santa Barbara Eyecare - Santa Barbara, Santa Barbara, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - ICON Eye Care - Grand Junction, Grand Junction, Colorado
  - Nature Coast Clinical Research - Crystal River, Crystal River, Florida
  - East Coast Institute for Research - Jacksonville, Jacksonville, Florida
  - Ocala Eye - 3130 Location, Ocala, Florida
  - Bascom Palmer Eye Institute - University of Miami Health System - Palm Beach Gardens, Palm Beach Gardens, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Coastal Research Associates, LLC. - Atlanta, Roswell, Georgia
  - Indiana University School of Medicine - Eugene and Marilyn Glick Eye Institute, Indianapolis, Indiana
  - Fraser Eye Care Center - Fraser, Fraser, Michigan
  - Great Lakes Eye Care - St. Joseph, Saint Joseph, Michigan
  - Huron Ophthalmology, P.C., Ypsilanti, Michigan
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - NV Eye Surgery - Henderson, Henderson, Nevada
  - Rochester Ophthalmological Group, PC - Brighton, Rochester, New York
  - "Clinic-LJ" Ltd, Winston-Salem, North Carolina
  - Cincinnati Eye Institute - Blue Ash, Cincinnati, Ohio
  - Abrams Eye Center, Inc., Cleveland, Ohio
  - AMA Eye Research Institute, Marysville, Ohio
  - Legacy Pulmonary Medical Group - Good Samaritan Medical Center, Portland, Oregon
  - Scott & White Cancer Center - Killeen, Cranberry Township, Pennsylvania
  - Scheie Eye Institute - University of Pennsylvania, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Advancing Vision Research - Goodlettsville, Goodlettsville, Tennessee
  - Total Eye Care, P.A., Memphis, Tennessee
  - Vanderbilt University Medical Center - Vanderbilt Eye Institute - Main Campus, Nashville, Tennessee
  - Texan Eye - Austin - Main Central, Austin, Texas
  - Southwest Eye Institute, El Paso, Texas
  - Houston Eye Associates - North Loop, Houston, Texas
  - Houston Eye Associates (HEA) - Gramercy Location, Houston, Texas
  - San Antonio Eye Center, P.A. - McCullough Ave, San Antonio, Texas
  - Rashid, Rice, Flynn & Reilly Eye Associates - San Antonio Clinic, San Antonio, Texas
  - St. George Eye Center - St. George, St. George, Utah
  - Piedmont Eye Center - Lynchburg, Lynchburg, Virginia
  - Specialty Eye Care Center - Bellevue, Bellevue, Washington
- Canada (2):
  - Prism Eye Institute - Oakville, Oakville, Ontario
  - Clinique Bellevue - Laval, Laval, Quebec
- Colombia (6):
  - Clínica Oftalmológica del Caribe, Barranquilla
  - Fundación Oftalmológica Nacional (FUNDONAL), Bogotá
  - Clinica de Oftalmologia de Cali SA, Cali
  - Fundación Oftalmológica de Santander FOSCAL, Floridablanca
  - Clinica de Oftalmologia Sandiego, Medellín
  - Instituto Nacional de Investigacion en Oftalmologia, Medellín